CLINICAL TRIAL: NCT02145234
Title: A Randomized, Placebo-Controlled, Single and Multiple Ascending Subcutaneous Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986089 in Healthy Adult Subjects
Brief Title: Placebo-Controlled, Single and Multiple Ascending Subcutaneous Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986089 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: CN001-001
Record Dates: First submitted 2014-05-16; First posted 2014-05-22 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- SAD Panel 1:BMS-986089/Placebo (Experimental): BMS-986089 in a single subcutaneous administration
  OR
  Placebo matching with BMS-986089 in a single subcutaneous administration
  Interventions: Drug: BMS-986089; Drug: Placebo matching with BMS-986089
- SAD Panel 2:BMS-986089/Placebo (Experimental): BMS-986089 in a single subcutaneous administration
  OR
  Placebo matching with BMS-986089 in a single subcutaneous administration
  Interventions: Drug: BMS-986089; Drug: Placebo matching with BMS-986089
- SAD Panel 3:BMS-986089/Placebo (Experimental): BMS-986089 in a single subcutaneous administration
  OR
  Placebo matching with BMS-986089 in a single subcutaneous administration
  Interventions: Drug: BMS-986089; Drug: Placebo matching with BMS-986089
- SAD Panel 4:BMS-986089/Placebo (Experimental): BMS-986089 in a single subcutaneous administration
  OR
  Placebo matching with BMS-986089 in a single subcutaneous administration
  Interventions: Drug: BMS-986089; Drug: Placebo matching with BMS-986089
- SAD Panel 5:BMS-986089/Placebo (Experimental): BMS-986089 in a single subcutaneous administration
  OR
  Placebo matching with BMS-986089 in a single subcutaneous administration
  Interventions: Drug: BMS-986089; Drug: Placebo matching with BMS-986089
- MAD Panel 1:BMS-986089/Placebo (Experimental): BMS-986089 in multiple subcutaneous administrations weekly
  OR
  Placebo matching with BMS-986089 multiple subcutaneous administrations weekly
  Interventions: Drug: BMS-986089; Drug: Placebo matching with BMS-986089
- MAD Panel 2:BMS-986089/Placebo (Experimental): BMS-986089 in multiple subcutaneous administrations weekly
  OR
  Placebo matching with BMS-986089 in multiple subcutaneous administrations weekly
  Interventions: Drug: BMS-986089; Drug: Placebo matching with BMS-986089
- MAD Panel 3:BMS-986089/Placebo (Experimental): BMS-986089 in multiple subcutaneous administrations weekly
  OR
  Placebo matching with BMS-986089 in multiple subcutaneous administrations weekly
  Interventions: Drug: BMS-986089; Drug: Placebo matching with BMS-986089
- MAD Panel 4:BMS-986089/Placebo (Experimental): BMS-986089 in multiple subcutaneous administrations weekly
  OR
  Placebo matching with BMS-986089 in multiple subcutaneous administrations weekly
  Interventions: Drug: BMS-986089; Drug: Placebo matching with BMS-986089
- MAD Panel 5:BMS-986089/Placebo (Experimental): BMS-986089 in multiple subcutaneous administration every 2 weeks
  OR
  Placebo matching with BMS-986089 in multiple subcutaneous administrations weekly
  Interventions: Drug: BMS-986089; Drug: Placebo matching with BMS-986089
- MAD Panel 6:BMS-986089/Placebo (Experimental): BMS-986089 in multiple subcutaneous administrations weekly
  OR
  Placebo matching with BMS-986089 in multiple subcutaneous administrations weekly
  Interventions: Drug: BMS-986089; Drug: Placebo matching with BMS-986089
- MAD Panel 7:BMS-986089/Placebo (Experimental): BMS-986089 a single subcutaneous administrations weekly
  OR
  Placebo matching with BMS-986089 a single subcutaneous administration every 2 weeks
  Interventions: Drug: BMS-986089; Drug: Placebo matching with BMS-986089

INTERVENTIONS:
Drug: BMS-986089
Drug: Placebo matching with BMS-986089

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, immunogenicity, pharmacokinetics and pharmacodynamics of single and multiple doses of BMS-986089 in healthy adult subjects.

DETAILED DESCRIPTION:
Primary Purpose - other: Protocol designed to assess the safety, tolerability, immunogenicity, Pharmacokinetics (PK) and Pharmacodynamics (PD) of BMS-986089 in healthy subjects

Enrollment: Single ascending dose panels: 48 subjects, Multiple ascending dose panels: 96

Minimum age: 18 years (Elderly MAD Panel 65 years of age) Maximum age: 55 years (Elderly MAD Panel 70 years of age)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal medical history, physical examination, ECGs and clinical laboratory determinations
* Men and women who are not of childbearing potential (ie, who are postmenopausal or Surgically sterile WOCBP) ages 21 to 55 years
* Women must not be breastfeeding
* Men who are sexually active with women of child bearing potential (WOCBP) must use any contraceptive method with a failure rate of less than 1% per year

Exclusion Criteria:

* Any significant acute or chronic medical illness Any major surgery within 6 weeks of study drug administration
* Any condition that will clearly require medical or surgical treatment during the period of study participation
* Any bone trauma or bone surgery within 3 months of study drug administration
* Known or suspected autoimmune disorder
* Donation of blood or plasma to a blood bank or in a clinical study (except at screening visit) within 6 weeks of study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Safety endpoints, including incidence of Adverse Event (AEs), serious AEs, AEs leading to discontinuation or death, as well as marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, and physical examinations | Single Ascending Dose (SAD) Phase 119 days
Safety endpoints, including incidence of Adverse Event (AEs), serious AEs, AEs leading to discontinuation or death, as well as marked abnormalities in clinical laboratory tests, vital sign measurements, ECGs, and physical examinations | Multiple Ascending Dose (MAD) phase 148 days

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) for SAD and MAD | SAD phase: Day1 to Day 91, MAD phase: Day 1 to Day 120
Time of maximum observed serum concentration (Tmax) for SAD and MAD | SAD phase: Day1 to Day 91, MAD phase: Day 1 to Day 120
Serum concentration 168 h post dose (C(168H)) for SAD and MAD | SAD phase: Day1 to Day 91, MAD phase: Day 1 to Day 120
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) for SAD | SAD phase: Day1 to Day 91
Area under the serum concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) for SAD | SAD phase: Day1 to Day 91
Apparent total body clearance (CLT/F) for SAD | SAD phase: Day1 to Day 91
Volume of distribution of terminal phase (if IV and if multi-exponential decline) (Vz/F) for SAD | SAD phase: Day1 to Day 91
Half life (T-Half) for SAD and MAD | SAD phase: Day1 to Day 91, MAD phase: Day 1 to Day 120
Serum concentration 336 h post dose (C(336H)) for SAD and MAD | SAD phase: Day1 to Day 91, MAD phase: Day 1 to Day 120
Effective elimination half-life that explains the degree of AUC accumulation observed (T-HALFeff_AUC) for MAD | MAD phase: Day 1 to Day 120
Area under the concentration-time curve in one dosing interval (AUC(TAU)) for MAD | MAD phase: Day 1 to Day 120
Degree of Fluctuation or Fluctuation Index (DF) for MAD | MAD phase: Day 1 to Day 120
Average concentration over a dosing interval (Css-Avg) for MAD | MAD phase: Day 1 to Day 120
AUC Accumulation Index; ratio of AUC(TAU) at steady state to AUC(TAU) after the first dose (AI AUC) for MAD | MAD phase: Day 1 to Day 120
Cmax Accumulation Index; ratio of Cmax at steady-state to Cmax after the first dose (AI Cmax) for MAD | MAD phase: Day 1 to Day 120
C(168H) Accumulation Index; ratio of C168H at steady-state to C168H after the first dose (AI C168H) for MAD | MAD phase: Day 1 to Day 120
C(336H) Accumulation Index; ratio of C(336H) at steady-state to C(336H) after the first dose (AI 336H) for MAD | MAD phase: Day 1 to Day 120
Immunogenicity of single and multiple doses of BMS-986089 will be measured by testing for the presence of ADAs for SAD and MAD | 30 days
The pharmacodynamic effect of single and multiple doses of BMS-986089 on free myostatin, total myostatin (pre-dose only), and myostatin-drug complex will be assessed by measuring these biomarkers for SAD and MAD | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Wcct Global, Llc, Cypress, California, United States

REFERENCES:
- [Derived] Muntoni F, Byrne BJ, McMillan HJ, Ryan MM, Wong BL, Dukart J, Bansal A, Cosson V, Dreghici R, Guridi M, Rabbia M, Staunton H, Tirucherai GS, Yen K, Yuan X, Wagner KR; Taldefgrobep Alfa Study Group. The Clinical Development of Taldefgrobep Alfa: An Anti-Myostatin Adnectin for the Treatment of Duchenne Muscular Dystrophy. Neurol Ther. 2024 Feb;13(1):183-219. doi: 10.1007/s40120-023-00570-w. Epub 2024 Jan 8. PMID 38190001
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx